CLINICAL TRIAL: NCT02236364
Title: Blood Glucose Monitoring Based on Imaging of the Eye
Brief Title: Noninvasive Blood Glucose Monitoring Method Based on Imaging of the Eye
Status: Terminated | Type: Observational
Why Stopped: The study was pulled by the sponsor due to lack of funding.
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: University of Toledo (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Other Study IDs: Irisense
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with type 1 or type 2 diabetes: Participants with type 1 or type 2 diabetes will have images of their iris collected at the same time as a fingerstick blood sugar
  Interventions: Device: Photographic Image Capture System

INTERVENTIONS:
Device: Photographic Image Capture System — Collection of images of the iris along with corresponding fingerstick blood glucose

SUMMARY:
Previous animal studies done by Dr. Brent Cameron in 2013 at the Univ. of Toledo have shown that glucose present in the fluid in the front of the eye, called the aqueous humor, correlates well with blood glucose. As blood glucose changes, the optical properties of the aqueous humor change, causing a change in the appearance of the iris of the eye.. The data collected in this study will be shared with IRISense to assist in validating the algorithm being used to develop the database needed. The data collected so far is in a narrow band of the normal glycemic range (healthy volunteers). We will collect standard digital photographic images of the eyes of subjects with diabetes along with corresponding blood glucose concentrations using the finger stick glucose monitoring method. In order to do this we will use standard digital photography techniques that is embedded in our benchtop prototype device

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diabetes Type 1 and 2 and can be verified by the principal investigator

Exclusion Criteria:

* Patients with any disease or abnormality of the eye
* Patients who are mentally incapacitated, cognitively impaired or with severe psychological disorders and cannot sign consent on their own

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetes Type 1 and 2
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- New Device for OPTICAL Determination of Blood Glucose Level: Single arm, using device to determine blood glucose level for all
Period: Overall Study
Arm/Group | New Device for OPTICAL Determination of Blood Glucose Level
Started | 25
Completed | 0
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | New Device for OPTICAL Determination of Blood Glucose Level
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 58.36 [23 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Data Acquisition for Continued Algorithm Development Using Photographic Images of the Iris Compared to Fingerstick Glucose Concentration
Description: Eight digital photographic image of the subject's iris will be obtained at various times during each visit under standard illumination using the developed instrumentation. A point-of-care fingerstick blood glucose reading will be taken with an FDA approved blood glucose measurement device (i.e., Contour, Bayer Healthcare, LLC) as close to simultaneously as possible with the photograph.
Time Frame: 60 day period
Population: The study was terminated by the sponsor prior to any analysis. Purpose of this study was to collect iris images for Sponsor's use in algorithm development. Images were stored in the prototype device that the Sponsor took back. Attempt was made to locate and contact the Sponsor, IRISense, but the company was dissolved in 2021. Since the company does not exist anymore neither does the data that the company was in possession of. Data is not available now nor will it be available in the future.
Arm/Group | New Device for OPTICAL Determination of Blood Glucose Level
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | New Device for OPTICAL Determination of Blood Glucose Level
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes